CLINICAL TRIAL: NCT01874015
Title: Transplantation of Bone Marrow Mesenchymal Stem Cell in Moderate to Severe Fistulizing Crohn's Disease
Brief Title: Transplantation of Bone Marrow Mesenchymal Stem Cell in Crohn's Disease
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Royan-GI-003
Record Dates: First submitted 2013-06-06; First posted 2013-06-10 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; mesenchymal stem cell; fistula
MeSH Terms: conditions — Crohn Disease; Fistula | interventions — Mesenchymal Stem Cell Transplantation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mesenchymal cell and fibroblast transplantaion (Active Comparator): The patients with crohn's disease who underwent mesenchymal cell and fibroblast injection.
  Interventions: Biological: mesenchymal cell and fibroblast injection
- mesenchymal cell transplantaion (Active Comparator): The patients with Crohn's disease who underwent mesenchymal cell transplantation.
  Interventions: Biological: mesenchymal cell transplantation

INTERVENTIONS:
Biological: mesenchymal cell transplantation — Mesenchymal cell transplantation in patients with Crohn's disease.
  Arms: mesenchymal cell transplantaion
Biological: mesenchymal cell and fibroblast injection — Transplantation of mesenchymal cell and fibroblast in patients with crohn's disease.
  Arms: mesenchymal cell and fibroblast transplantaion

SUMMARY:
This study is a prospective, randomized, parallel, phase 1 trial to assess the safety and feasibility of the transplantation of bone marrow derived mesenchymal stem cells (MSCs) in fistulizing Crohn's disease.

DETAILED DESCRIPTION:
In this study all eligible patients were randomly allocated into two study groups by a permuted block randomization method: group A receives only autologous MSCs suspended in fibrin glue, group B receives autologous MSCs+ Fibroblasts. Both groups receive 4 injections inside the wall and lumen of the fistula. Injections will be repeated every month.

ELIGIBILITY:
Inclusion Criteria:

* 1- Poor response to routine treatments in refractory Crohn's disease with fistula.

  2- CDAI>220 3- Age 18 to 60 years 4- GFR>30, Cr<2 5- The presence of perinea fistula.

Exclusion Criteria:

* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-02 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
fistula closure | 4months
  Evaluation the fistula closure after mesenchymal cell transplantation in patients with crohn's disease.

SECONDARY OUTCOMES:
CDAI | 4months
  Evaluation the decrease of CDAI after mesenchymal cell transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Nasser Aghdami, MD,PhD, Study Director — Head of Royan department of degenerative medicine,Head of Royan celltherapy center; Mahdi Mohammad Nejhad, MD, Study Director — TUMS DDRI
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- See also: Related Info — http://Royaninstitute.org